CLINICAL TRIAL: NCT01737034
Title: Ätiologie, Pathophysiologie Und Prävention Einer überschießenden Körperfettzunahme Nach Gewichtsreduktion - Vermeidung Des JoJo-Effektes in Der Behandlung Von Übergewicht
Brief Title: A Low Glycemic Index Diet as Prevention of the Catch-up Fat Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Manfred James Müller, Principal Investigator, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMBF 0315681
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Dietary Intervention
Keywords: partitioning of weight gain; refeeding; catch-up fat phenomenon; glycemic index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- low GI, low GI (Experimental): low GI diet (semi starvation phase) followed by low GI diet in the refeeding phase
  Interventions: Other: dietary intervention by varying GI diets
- low GI, high GI (Experimental): low GI diet (semi starvation phase) followed by high GI diet in the refeeding phase
  Interventions: Other: dietary intervention by varying GI diets
- high GI, low GI (Experimental): high GI diet (semi starvation phase) followed by low GI diet in the refeeding phase
  Interventions: Other: dietary intervention by varying GI diets
- high GI, high GI (Experimental): high GI diet (semi starvation phase) followed by high GI diet in the refeeding phase
  Interventions: Other: dietary intervention by varying GI diets

INTERVENTIONS:
Other: dietary intervention by varying GI diets — The human study intends to characterise the partitioning of weight gain during refeeding and to affect the catch-up fat phenomenon by the glycemic index (GI) of the diet.

SUMMARY:
The catch-up fat phenomenon is an evolutionary conserved physiological response to a starvationrefeeding cycle. It is characterized by long-term suppression of thermogenesis, reduced body protein regain and an increase in fat mass above basal level during refeeding. Clinically, it characterises weight cycling in overweight patients which is associated with increasing fat mass (visceral fat) and increased morbidity (e.g. insulin resistance, inflammation). In this project, the physiological, cellular and molecular mechanisms of this phenomenon will be investigated in humans, mice and C. elegans. It is hypothesized that refeeding a low GI (=glycemic index)- diet after weight loss prevents the catchup fat phenomenon and its sequelae. This translational research will provide comprehensive insights into the catch-up fat phenomenon as well as provide a suitable strategy of its prevention.

DETAILED DESCRIPTION:
In a human intervention study, changes in physiological, metabolic, and neuroendocrine functions in response to weight cycling will be investigated under controlled conditions in normal weight subjects. The mechanisms of the catch-up fat phenomenon are analysed starting from stable energy balance followed by overfeeding, weight loss and weight regain following weight loss (refeeding). Changes in body composition (including ectopic fat), metabolism (resting energy expenditure, substrate oxidation rates, insulin resistance) and plasma hormone concentrations will be assessed. Fat tissue probes will be used to characterise key enzymes and signalling pathways, redox status and whole genome expression. Modulation of the hormonal response to weight cycling is brought about by varying macronutrient content and glycemic index of the diets. We hypothesize that, insulin and leptin resistance are explained by increased insulin secretion during the refeeding period. Both, adaptive thermogenesis as well as insulin and leptin resistance can be ameliorated by attenuation of the increase in insulin and leptin secretion during refeeding a low GI diet after weight loss.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (BMI 20-24 kg/m2), normal fat mass

Exclusion Criteria:

* smoking, chronic diseases, drug intake, nutrient allergies, lactose intolerance, pacemaker, metalliferous implants

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in body composition and energy metabolism after 3 weeks of underfeeding and 2 following weeks of refeeding | Body composition measurement after 4 and 6 study weeks
  Body composition measurement including BODPOD, QMR, BIA Energy Metabolism measurement using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Manfred J. Müller, Prof., Study Chair — Institute of Human Nutrition, University of Kiel
Locations (1):
- Institute of Human Nutrition, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Breusing N, Lagerpusch M, Engstler AJ, Bergheim I, Mueller MJ, Bosy-Westphal A. Influence of Energy Balance and Glycemic Index on Metabolic Endotoxemia in Healthy Men. J Am Coll Nutr. 2017 Jan;36(1):72-79. doi: 10.1080/07315724.2016.1156036. Epub 2017 Jan 6. PMID 28060600
- [Derived] Geisler C, Braun W, Pourhassan M, Schweitzer L, Gluer CC, Bosy-Westphal A, Muller MJ. Gender-Specific Associations in Age-Related Changes in Resting Energy Expenditure (REE) and MRI Measured Body Composition in Healthy Caucasians. J Gerontol A Biol Sci Med Sci. 2016 Jul;71(7):941-6. doi: 10.1093/gerona/glv211. Epub 2015 Nov 20. PMID 26590912
- [Derived] Muller MJ, Enderle J, Pourhassan M, Braun W, Eggeling B, Lagerpusch M, Gluer CC, Kehayias JJ, Kiosz D, Bosy-Westphal A. Metabolic adaptation to caloric restriction and subsequent refeeding: the Minnesota Starvation Experiment revisited. Am J Clin Nutr. 2015 Oct;102(4):807-19. doi: 10.3945/ajcn.115.109173. Epub 2015 Sep 23. PMID 26399868
- [Derived] Schweitzer L, Geisler C, Pourhassan M, Braun W, Gluer CC, Bosy-Westphal A, Muller MJ. What is the best reference site for a single MRI slice to assess whole-body skeletal muscle and adipose tissue volumes in healthy adults? Am J Clin Nutr. 2015 Jul;102(1):58-65. doi: 10.3945/ajcn.115.111203. Epub 2015 May 27. PMID 26016860
- [Derived] Karschin J, Lagerpusch M, Enderle J, Eggeling B, Muller MJ, Bosy-Westphal A. Endocrine determinants of changes in insulin sensitivity and insulin secretion during a weight cycle in healthy men. PLoS One. 2015 Feb 27;10(2):e0117865. doi: 10.1371/journal.pone.0117865. eCollection 2015. PMID 25723719
- [Derived] Lagerpusch M, Enderle J, Eggeling B, Braun W, Johannsen M, Pape D, Muller MJ, Bosy-Westphal A. Carbohydrate quality and quantity affect glucose and lipid metabolism during weight regain in healthy men. J Nutr. 2013 Oct;143(10):1593-601. doi: 10.3945/jn.113.179390. Epub 2013 Aug 14. PMID 23946346